CLINICAL TRIAL: NCT04109209
Title: NeuroCARE: Psychological Intervention for Caregivers of Patients With Malignant Gliomas (RCT)
Brief Title: Psychological Intervention For Brain Tumor Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Principal Investigator, Deborah A Forst, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 19-250
Record Dates: First submitted 2019-09-26; First posted 2019-09-30 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Malignant Glioma; Anxiety; Caregiver Burden; Malignant Brain Tumor
Keywords: Malignant Glioma; Caregiver Anxiety; Caregiver Burden; Psychological distress; Brain Tumor
MeSH Terms: conditions — Glioma; Anxiety Disorders; Caregiver Burden; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care Group (Active Comparator): * 60 Participants will be randomized to receive usual care for caregivers of patients with malignant brain tumors
  * Caregivers randomized to the usual care arm will be referred to the brain tumor clinic social worker or other appropriate cancer center resources upon request from the caregiver, patient or clinician
  * Complete 3 questionnaires: Baseline, 11 weeks, 16 weeks
  Interventions: Behavioral: Usual Care Group
- Psychosocial Intervention Group (Experimental): * 60 Participants of caregivers of patients with malignant brain tumors will be randomized into the psychosocial intervention arm
  * Caregivers assigned to the intervention arm will receive usual care and the psychosocial intervention. The intervention entails six one-on-one sessions with an interventionist (psychologist or social worker)
  * Complete 3 questionnaires: Baseline, 11 weeks, 16 weeks
  Interventions: Behavioral: Psychosocial Intervention Group

INTERVENTIONS:
Behavioral: Psychosocial Intervention Group — The intervention will consist of six one-on-one sessions (45 minutes each). Complete 3 questionnaires: Baseline, 11 weeks, 16 weeks
  Arms: Psychosocial Intervention Group
Behavioral: Usual Care Group — Caregivers randomized to the usual care arm will be referred to the brain tumor clinic social worker or other appropriate cancer center resources upon request from the caregiver, patient or clinician
  •Complete 3 questionnaires: Baseline, 11 weeks, 16 weeks
  Arms: Usual Care Group

SUMMARY:
This study is testing a supportive psychosocial intervention for caregivers of people who have malignant brain tumors such as gliomas or other high-grade primary brain tumors. This study was designed because caregivers of patients with malignant brain tumors often experience physical and psychological burdens caring for their loved ones.

The purpose of this study is to find out whether a program offering psychological support can help caregivers learn effective coping methods during their loved one's treatment and make the experience of being a caregiver more manageable.

DETAILED DESCRIPTION:
This study will be a prospective, randomized controlled trial to assess the efficacy of a caregiver-directed intervention designed to improve anxiety in caregivers of patients with malignant brain tumors, in comparison with caregivers who receive usual care.

The aim of this study is to test the efficacy of this intervention in reducing distress in caregivers of patients with malignant brain tumors, in comparison with usual care. The study will be conducted in 120 caregivers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Identified by study staff, a clinician, self, or a patient with a malignant brain tumor as the patient's primary caregiver
* The patient is receiving care at the MGH Cancer Center
* The patient was diagnosed with a malignant brain tumor within the past 6 months
* Able to speak and read in English
* Generalized Anxiety Disorder 7-item (GAD-7) score ≥5
* Participants may or may not be pregnant.

Exclusion Criteria:

* Deemed inappropriate for the study by the patient's clinician or the study PI
* Participated in the pilot study of this caregiver intervention (DF/HCC 18-426)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2019-10-09 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
Anxiety symptoms | 11 weeks
  We will compare anxiety symptoms using the Anxiety Subscale of the Hospital Anxiety and Depression Scale (HADS-A) between the intervention and usual care group. The HADS-A is a 7-item subscale with scores ranging from 0 to 21, with higher scores indicating higher levels of anxiety.

SECONDARY OUTCOMES:
Anxiety symptoms longitudinally | Up to 16 weeks
  We will compare anxiety symptoms using the Anxiety subscale of the hospital anxiety and depression scale (HADS-A) between the two groups longitudinally. HADS-A is the 7-item anxiety subscale of the Hospital Anxiety and Depression Scale. Scores range from 0 to 21, with higher scores indicating higher levels of anxiety.
Self-Efficacy | Up to 16 weeks
  Comparison of the effect of the intervention on caregiver self-efficacy (CASE) between study groups . The Lewis Cancer Self-Efficacy Scale (CASE) is a 17-item scale that measures caregivers' confidence in managing the impact of their loved one's illness from. Score range from 0 to 170. Higher scores indicate higher self-efficacy.
Coping skills | Up to 16 weeks
  We will compare coping skills between study arms using the Measure of Current Status Part A (MOCS-A). The MOCS-A assesses caregivers' self-perceived status on coping skills targeted by the intervention. Total MOCS-A scores range from 0-52 with higher scores indicating better self-perceived coping skills.
Quality of life using the Caregiver quality of life oncology questionnaire | Up to 16 weeks
  Comparison of caregiver quality of life (CarGOQoL) between study groups. The CareGiver Oncology QoL questionnaire (CarGOQoL) is a 29-item, well-validated instrument specific to caregivers for patients with cancer, used to measure family caregiver QoL in multiple domains. Overall scores range from 0 to 100, with higher scores corresponding to higher quality of life.
Caregiver burden | Up to 16 weeks
  Comparison of caregiver burden (CRA) between study groups.
  - Caregiving burden will be measured using the Caregiver Reaction Assessment (CRA), a 24-item scale measuring caregiving burden with score range of 24-120. Higher scores indicate higher caregiving burden.
Depression symptoms | Up to 16 weeks
  Comparison of the effect of the intervention on depression symptoms (HADS-D) between study groups. HADS-D is the 7-item depression subscale of the Hospital Anxiety and Depression Scale. Scores range from 0 to 21, with higher scores indicating higher levels of depression.
PTSD symptoms | Up to 16 weeks
  Comparison of post-traumatic stress disorder (PTSD) symptoms between study groups . PTSD symptoms will be measured using the PCL-5, a 20-item questionnaire with scores ranging from 0-80; higher scores indicate more severe PTSD symptoms.

OTHER OUTCOMES:
Intervention Acceptability | 11 weeks
  For participants who are assigned to the intervention arm, we will use the Client Satisfaction Questionnaire (CSQ-3), a three-item questionnaire designed to evaluate satisfaction with provision, quality, and outcome of services, to assess participant acceptability of the NeuroCARE intervention. Total scores on the CSQ-3 range from 4-12, with higher numbers indicating a higher level of satisfaction with the services provided.
Exploratory Moderation Analysis | Up to 16 weeks
  As an exploratory analysis, we will assess whether age, sex, and baseline anxiety moderate the effect of the intervention on caregiver reported outcomes
Exploratory Causal Mediation Analysis | Up to 16 weeks
  Exploratory causal mediation analysis to explore whether caregiver self-efficacy and coping skills mediate the effect of the intervention on caregiver anxiety symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Deborah Forst, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] Forst DA, Podgurski AF, Strander SM, Whitman JD, Datta S, Pintro K, Horick NK, Willis KD, Sannes TS, Greer JA, El-Jawahri A, Jacobs JM, Temel JS. NeuroCARE: A Randomized Controlled Trial of a Psychological Intervention for Caregivers of Patients With Primary Malignant Brain Tumors. J Clin Oncol. 2024 Dec 20;42(36):4252-4262. doi: 10.1200/JCO.24.00065. Epub 2024 Sep 16. PMID 39284103
- [Derived] Forst DA, Rhee JY, Mesa MM, Podgurski AF, Strander SM, Datta S, Kaslow-Zieve E, Horick NK, Greer JA, El-Jawahri A, Sannes TS, Temel JS, Jacobs J. Study protocol for NeuroCARE: a randomised controlled trial of a psychological intervention for caregivers of patients with primary malignant brain tumours. BMJ Open. 2023 Sep 7;13(9):e069410. doi: 10.1136/bmjopen-2022-069410. PMID 37678946